CLINICAL TRIAL: NCT05254353
Title: Comparison of Different CSF Sampling Sites on External Ventricular Drains
Acronym: CSF3S
Status: Recruiting | Type: Observational
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Sponsor
Other Study IDs: S65845
Record Dates: First submitted 2022-01-19; First posted 2022-02-24 (Actual); Last update posted 2024-07-01 (Actual); Status verified 2024-06

CONDITIONS: Cerebrospinal Fluid
Keywords: neurosurgery; CSF; EVD

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — CSF
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with EVD
  Interventions: Procedure: Analyses of proximal and distal samples

INTERVENTIONS:
Procedure: Analyses of proximal and distal samples — Evaluate the difference between proximal and distal CSF samples

SUMMARY:
The aim of the current study is to evaluate the difference between proximal and distal CSF sampling. If the characteristics of distally and proximally sampled CSF are similar or correlate well, it may be possible to only sample CSF distally in the future, thereby avoiding the risks mentioned above.

DETAILED DESCRIPTION:
Insertion of an external ventricular drain (EVD) is a common neurosurgical procedure, for example in patients with intracranial bleeding, head trauma of tumours. The aim of an external ventricular drain is either to drain cerebrospinal fluid (CSF) or to measure intracranial pressure. In patients with external ventricular drains, it is a common practice in many centres, including UZ Leuven, to routinely sample CSF two or three times a week. The following tests are routinely performed: protein level, glucose level, lactate level, white cell count, red cell count, and cultures. Gram stain is performed in case white blood cell count exceeds 5 cells/mm³. This regular sampling (1) permits early detection of ventriculitis, which may be rather asymptomatic, especially in sedated patients,and (2) may guide neurosurgeons to the ideal timeframe to either taper the external ventricular drainage, or replace it by a ventriculoperitoneal shunt.

A typical external ventricular drainage system consists of a ventricular catheter, which is nowadays usually impregnated with antibiotics (e.g. Codman Bactiseal - coated with clindamycin and rifampicin), an extension tube, a drip chamber, and a collection bag. Multiple three-way taps and access ports along its course allow for CSF sampling (or injection of therapeutics, such as tissue plasminogen activator, or saline to flush the catheter in case of blockage).

From a practical perspective, CSF sampling from the external ventricular drain is possible at all of these three-way taps and access ports. Broadly, one may sample CSF as proximally (close to the ventricle) as possible (e.g. by using the access port), or distally (at the level of the drip chamber, e.g. by using the three-way tap between the drip chamber and the collection bag). There is no consistency in for CSF collection site amongst different institutions. Traditionally, in UZ Leuven, we have been sampling CSF proximally until now.

The main theoretical advantage of proximal sampling is that actively aspirated "fresh" CSF close to the ventricle likely closely resembles the true characteristics of our study object, i.e. intraventricular CSF. Nevertheless, this approach is not without risk. First, it requires to directly access the sterile inside of the extension tube. This inherently comes with a risk of iatrogenic infection. Secondly, by aspirating the external ventricular catheter, the neurosurgeon may induce an iatrogenic haemorrhage in the brain parenchyma or the ventricle, and/or direct trauma to the brain parenchyma, as in suboptimally positioned catheters or small ventricles, white matter or choroid plexus may be aspirated along with CSF. Because of the risk of iatrogenic infections, haemorrhage or trauma, it is our institutional policy that CSF sampling from external ventricular drains is performed by neurosurgeons only. This also poses practical problems and may delay sampling, especially in patients who are not admitted to neurosurgical wards (e.g. paediatric cases).

From a theoretical perspective, distal CSF sampling, at the level of the drip chamber, has multiple advantages. First, the risk of iatrogenic infections induced by CSF sampling is likely to be lower, as there is no direct contact between the CSF in the drip chamber and the intraventricular CSF. Secondly, there is no risk of inducing haemorrhages or brain trauma, as no "active" aspiration is required for CSF sampling. Hence, distal CSF sampling can perhaps also be carried out by physicians from other fields than neurosurgery, or by trained nurses. However, theoretically, it is possible that the characteristics of CSF sampled distally do not sufficiently resemble those of intraventricular CSF.

ELIGIBILITY:
Inclusion Criteria:

* Patients with an EVD in place regardless of the underlying pathology.
* Written informed consent to participate in the study must be obtained from the subject. If the subject is not capable of self-consent, all efforts will be made to locate a legally acceptable representative to act on behalf of the subject.

When the patient is considered capable to consent but physically unable to sign an informed consent form and a representative is not available an impartial witness can attend the informed consent process.

- Males and females of all ages, including children and pregnant females

Exclusion Criteria:

* Patients in whom the removal of the drain is planned within 48 hours, before routine sampling, will be excluded.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with an external ventricular drain (EVD) presenting to the Neurosurgery ward.
Sampling Method: Probability Sample
Enrollment: 55 (Estimated)
Dates: Start 2022-01-31 (Actual); Primary Completion 2025-01 (Estimated); Study Completion 2025-01 (Estimated)

PRIMARY OUTCOMES:
Change of the CSF white cell count at day 1-4 and day 5-9 when comparing both sampling methods | Day 1-4 and day 5-9 after placement of EVD
  The aim of the current study is to evaluate the difference between proximal and distal CSF sampling.

SECONDARY OUTCOMES:
White cell count correlation for all the available time points | Samples will be taken every 2-3 days after placement until removal of EVD (estimated between 7 and 28 days)
Gram stain correlation for all the available time points | Samples will be taken every 2-3 days after placement until removal of EVD (estimated between 7 and 28 days)
Culture correlation for all the available time points | Samples will be taken every 2-3 days after placement until removal of EVD (estimated between 7 and 28 days)
Protein correlation for all the available time points | Samples will be taken every 2-3 days after placement until removal of EVD (estimated between 7 and 28 days)
Glucose correlation for all the available time points | Samples will be taken every 2-3 days after placement until removal of EVD (estimated between 7 and 28 days)
Lactate correlation for all the available time points | Samples will be taken every 2-3 days after placement until removal of EVD (estimated between 7 and 28 days)
Red cell count correlation for all the available time points | Samples will be taken every 2-3 days after placement until removal of EVD (estimated between 7 and 28 days)
Absolute difference between white blood cell count, protein, glucose, lactate, and red blood cell count | Samples will be taken every 2-3 days after placement until removal of EVD (estimated between 7 and 28 days)
AEs likely related to CSF sampling, irrespective of the method (new or increased haemorrhage, infection) | Samples will be taken every 2-3 days after placement until removal of EVD (estimated between 7 and 28 days)

CONTACTS AND LOCATIONS:
Overall Officials: Philippe De Vloo, prof.dr., Principal Investigator — UZ Leuven
Locations (1):
- UZ Leuven, Leuven, Belgium